CLINICAL TRIAL: NCT01436968
Title: A Randomized Controlled Trial of ProstAtak® as Adjuvant to Up-front Radiation Therapy For Localized Prostate Cancer
Brief Title: Phase 3 Study of ProstAtak® Immunotherapy With Standard Radiation Therapy for Localized Prostate Cancer
Acronym: PrTK03
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Candel Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PrTK03
Record Dates: First submitted 2011-09-19; First posted 2011-09-20 (Estimated); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Prostate Cancer
Keywords: immunotherapy, cytotoxicity, tumor vaccine, prostate cancer, radiotherapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Valacyclovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ProstAtak® (Experimental): Aglatimagene besadenovec (CAN-2409) + valacyclovir + radiation therapy +/- ADT
  Interventions: Biological: Aglatimagene besadenovec + valacyclovir
- Control (Placebo Comparator): Placebo + valacyclovir + radiation therapy +/- ADT
  Interventions: Biological: Placebo + valacyclovir

INTERVENTIONS:
Biological: Aglatimagene besadenovec + valacyclovir — Patients will receive three courses of ProstAtak® each consisting of aglatimagene besadenovec injection + oral valacyclovir. AdV-tk injection will be delivered to the prostate via trans-rectal ultrasound guided injection as follows:
  1. The first injection will be given at least 15 days and not more than 8 weeks before starting radiation.
  2. The second injection will be 0-3 days before initiation of radiation therapy.
  3. The third injection will be 15-22 days after the 2nd injection.
  The prodrug, valacyclovir, will be administered at a fixed dose for 14 days after each AdV-tk injection.
  Standard external beam radiation therapy will be delivered to the prostate. Short-term androgen deprivation therapy (maximum of 6 months) is optional but must be decided before enrollment to allow for stratification.
  Other Names: AdV-tk; CAN-2409
  Arms: ProstAtak®
Biological: Placebo + valacyclovir — Patients will receive three courses each consisting of placebo injection + oral valacyclovir. Placebo injection will be delivered to the prostate via trans-rectal ultrasound guided injection as follows:
  1. The first injection will be given at least 15 days and not more than 8 weeks before starting radiation.
  2. The second injection will be 0-3 days before initiation of radiation therapy.
  3. The third injection will be 15-22 days after the 2nd injection.
  The prodrug, valacyclovir, will be administered at a fixed dose for 14 days after each placebo injection.
  Standard external beam radiation therapy will be delivered to the prostate. Short-term androgen deprivation therapy (maximum of 6 months) is optional but must be decided before enrollment to allow for stratification.
  Arms: Control

SUMMARY:
The purpose of this study is to evaluate the effectiveness of ProstAtak® immunotherapy in combination with radiation therapy for patients with intermediate-high risk localized prostate cancer. ProstAtak kills tumor cells and stimulates a cancer vaccine effect. Killing tumor cells in an immune stimulatory environment induces the body's immune system to detect and destroy cancer cells. ProstAtak has shown synergy with radiation without added toxicity and lower than expected recurrence rates in previous clinical trials. The hypothesis is that ProstAtak can lead to improvement in the clinical outcome for patients with prostate cancer. Participants will be randomized to the ProstAtak or control arm at a 2:1 ratio. Both arms receive standard external beam radiation therapy. Short-term androgen deprivation therapy may be given but is not required.

ELIGIBILITY:
Inclusion Criteria include:

* Localized prostate cancer meeting the NCCN criteria of Intermediate Risk or patients having only one NCCN high-risk feature

  * NCCN Intermediate Risk is defined as having at least one of the following: PSA 10-20 ng/ml, Gleason score =7, T2b-T2c
  * High Risk with a single high risk feature is defined as having only one of the following: PSA>20 ng/ml, Gleason score 8-10, or T3a
  * Excluded are those in the following risk groups: Low risk; High risk with more than 1 high risk factor; Locally advanced/very high risk=T3b-T4; Metastatic: N1 or M1
* Planning to undergo standard prostate-only external beam radiation therapy
* ECOG Performance Status 0-2

Exclusion Criteria include:

* Liver disease, including known cirrhosis or active hepatitis
* Patients on systemic corticosteroids (>10mg prednisone per day) or other immunosuppressive drugs
* Known HIV+ patients
* Regional lymph node involvement or distant metastases
* Patients planning to receive whole pelvic irradiation
* Prior treatment for prostate cancer, except TURP or ADT. For ADT, it may only be given for a maximum of 6 months
* Patients who had or plan to have orchiectomy as the form of hormonal ablation
* Known sensitivity or allergic reactions to acyclovir or valacyclovir

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 711 (Estimated)
Dates: Start 2011-09; Primary Completion 2024-08 (Actual); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Disease free survival defined as the time from randomization until the date of the first failure event will be compared for the ProstAtak® arm versus the placebo control arm. The analyses will be based on the intent to treat population. | Assessed at each visit every 6 months through year 5 until event occurs.

SECONDARY OUTCOMES:
Prostate cancer specific survival and overall survival will be compared for the ProstAtak® arm versus the placebo control arm. | Assessed at each visit every 6 months through year 5 after which long-term follow up of general health status will continue yearly.
PSA nadir will be compared for the ProstAtak® arm versus the placebo control arm. | Assessed at each visit every 6 months through year 5.
Patient reported Health Related Quality of Life outcomes will be collected using the Expanded Prostate Cancer Index Composite (EPIC-26) questionnaire. The change in QOL over time will be compared for the ProstAtak® arm versus the placebo control arm. | Assessed at baseline and at 3, 6, 12, 18 and 24 months after completion of radiation.
The safety profile will be characterized by collection of adverse event information and laboratory values during the treatment phase (until the completion of radiation). Data on late effects will be collected after radiation completion. | Assessed at each visit and continuously throughout the study.

CONTACTS AND LOCATIONS:
Locations (73):
- United States (72):
  - Arizona Center for Cancer Care - Gilbert, Gilbert, Arizona
  - Arizona Urology Specialists, Glendale, Arizona
  - Arizona Oncology Services Foundation, Multiple Locations, Arizona
  - Arizona Center for Cancer Care - Peoria, Peoria, Arizona
  - Arizona Center for Cancer Care - Deer Valley, Phoenix, Arizona
  - Arizona Center for Cancer Care - Osborne, Scottsdale, Arizona
  - Arizona Center for Cancer Care - Shea, Scottsdale, Arizona
  - Arizona Center for Cancer Care - Surprise, Surprise, Arizona
  - Southern Arizona VA Health Care System, Tucson, Arizona
  - VA Northern California Health Care System, Mather, California
  - Precision Radiation Oncology, Tustin, California
  - Valley View Hospital, Glenwood Springs, Colorado
  - Colorado Clinical Research, Lakewood, Colorado
  - Advanced Urology, Parker, Colorado
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - 21st Century Oncology, Fort Lauderdale, Florida
  - 21st Century Oncology, Lakewood Rch, Florida
  - 21st Century Oncology, Naples, Florida
  - 21st Century Oncology, Plantation, Florida
  - Clinical Research Center of Florida, Pompano Beach, Florida
  - James A. Haley Veteran's Hospital, Tampa, Florida
  - Florida Urology Partners, Tampa, Florida
  - Jesse Brown VA Medical Center, Chicago, Illinois
  - The University of Chicago, Chicago, Illinois
  - Silver Cross Hospital, New Lenox, Illinois
  - Southeast Louisiana Veterans Health Care System, New Orleans, Louisiana
  - VA Maryland Health Care System, Baltimore, Maryland
  - Chesapeake Urology Research Associates, Baltimore, Maryland
  - The Johns Hopkins University School of Medicine, The Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Kansas City VA Medical Center, Kansas City, Missouri
  - Adult & Pediatric Urology, P.C., Omaha, Nebraska
  - Sheldon Freedman MD, Ltd., Las Vegas, Nevada
  - VA Sierra Nevada Health Care System, Reno, Nevada
  - New Jersey Urology - Cherry Hill, Cherry Hill, New Jersey
  - New Jersey Urology - Englewood, Englewood, New Jersey
  - New Jersey Urology - Milburn, Millburn, New Jersey
  - New Jersey Urology - Saddle Brook, Saddle Brook, New Jersey
  - New Jersey Urology - West Orange, West Orange, New Jersey
  - New Mexico Oncology Hematology Consultants (NMOHC), Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Advanced Radiation Centers of New York (Integrated Medical Professionals), North Hills, New York
  - Associated Medical Professionals of NY, PLLC, Syracuse, New York
  - James J. Peters VA Medical Center, The Bronx, New York
  - Durham VA Health Care System, Durham, North Carolina
  - Cincinnati VA Medical Center, Cincinnati, Ohio
  - VA Portland Health Care System, Portland, Oregon
  - Oregon Urology Institute, Springfield, Oregon
  - MidLantic Urology, Bala-Cynwyd, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Ralph H. Johnson Veterans Affairs Medical Center, Charleston, South Carolina
  - Carolina Urologic Research Center, LLC, Myrtle Beach, South Carolina
  - Urology Austin, Austin, Texas
  - Austin Urology Institute, Austin, Texas
  - Austin Urology Institute - Northwest Austin Cancer Center, Austin, Texas
  - VA North Texas Health Care System, Dallas, Texas
  - Urology Clinics of North Texas, Dallas, Texas
  - Dr. Irving Fishman's Office, Houston, Texas
  - Houston Willowbrook Radiation Oncology, Houston, Texas
  - Dr. Ned Stein's Office, Houston, Texas
  - South Texas San Antonio VA Healthcare System, San Antonio, Texas
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Texas Urology Specialists-The Woodlands, The Woodlands, Texas
  - The Methodist Hospital - The Woodlands, The Woodlands, Texas
  - Texas Urology Specialists, Tomball, Texas
  - Potomac Urology Center, Alexandria, Virginia
  - Hunter Holmes McGuire VA Medical Center, Richmond, Virginia
  - Salem VA Medical Center, Salem, Virginia
  - Urology of Virginia, PLLC, Virginia Beach, Virginia
  - MultiCare Regional Cancer Center - Gig Harbor, Gig Harbor, Washington
  - MultiCare Regional Cancer Center - Tacoma, Tacoma, Washington
- VA Caribbean Healthcare System, San Juan, Puerto Rico